CLINICAL TRIAL: NCT05088278
Title: Long Term Clinical and Radiographical Outcomes of Different Anterior Cruciate Ligament Reconstruction Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Long term ACLR
Record Dates: First submitted 2021-10-12; First posted 2021-10-21 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Anterior Cruciate Ligament Tear; Osteoarthritis, Knee
Keywords: anterior cruciate ligament; knee osteoarthritis; hamstrings; patellar tendon; lateral extra articular tenodesis
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HS (Active Comparator): Patients who underwent anatomical single-bundle ACL reconstruction with hamstrings
  Interventions: Procedure: Anatomical single bundle ACL reconstruction with hamstrings
- BPT (Active Comparator): Patients who underwent anatomical single-bundle ACL reconstruction with patellar tendon
  Interventions: Procedure: Anatomical single bundle ACL reconstruction with patellar tendon
- Over-the-top plus lateral plasty (Experimental): Patients who underwent ACL reconstruction with Over-the-top plus lateral plasty technique
  Interventions: Procedure: ACL reconstruction with over the top plus lateral plasty technique

INTERVENTIONS:
Procedure: Anatomical single bundle ACL reconstruction with hamstrings — Anatomical ACL reconstruction with quadruple-bundle hamstrings graft
  Arms: HS
Procedure: Anatomical single bundle ACL reconstruction with patellar tendon — Anatomical single bundle ACL reconstruction with patellar tendon
  Arms: BPT
Procedure: ACL reconstruction with over the top plus lateral plasty technique — Non-anatomical ACL reconstruction, the hamstrings' tibial insertion is preserved; a double-bundle hamstring graft is passed intra-articularly, fixed in over the top position on the lateral femoral condyle, and then passed extra-articularly deeply to ileo-tibial band up to the tibia, where it is fixed at the level of Gerdy's tubercle.
  Arms: Over-the-top plus lateral plasty

SUMMARY:
The purpose of this study is to evaluate the long-term results of various anterior cruciate ligament reconstruction techniques. This assessment is necessary for the current context of anterior cruciate ligament research as several techniques and grafts are used in clinical practice, however, the various studies existing in the literature focus mainly only on the direct comparison of two techniques and usually with short-to-medium term follow-up. Since gonarthrosis is one of the most debated consequences of cruciate ligament reconstruction, a comparison of different long-term procedures would be desirable to have a clearer picture of the risks and benefits associated with different types of intervention.

DETAILED DESCRIPTION:
In the beginning, the Database of our Institute is consulted, all the patients that underwent ACL reconstruction at least 15 years ago are selected. The original group will be divided into subgroups based on the surgical technique adopted, of the different techniques we took into consideration only these three: anatomical ACL reconstruction with patellar tendon, anatomical ACL reconstruction with hamstrings, non-anatomical ACL reconstruction "Over-the-top plus lateral plasty". The patients will be contacted to ask if they are interested to take part in the study; at least 25 patients for each group will be recruited. All the patients recruited will sign an informed consent about the study and the personal data treatment. After consent acquisition, patients will undergo a clinical examination and a questionnaire about pain and knee status will be administered; moreover, a radiographical examination of the operated knee will be performed to assess the osteoarthritis progression. Patients that reported graft rupture will be registered as failures.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent ACL reconstruction with single-bundle anatomical technique (patellar tendon, semitendinous and gracile tendons) or "Over-The-Top plus lateral plastic" technique and any associated procedures with at least 15 years of follow up;
2. Patients aged between 15 and 50 at the time of surgery;
3. Patients with isolated ACL tear;
4. Patients with healthy contralateral knee at the time of surgery.

Exclusion Criteria:

1. Patients with grade III-IV chondral lesions according to Outerbridge scale at surgery;
2. Patients no longer available;
3. Women of childbearing age who cannot exclude pregnancy;
4. Patients unable to give informed consent or patients unwilling to sign informed consent.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-07-27 (Actual)

PRIMARY OUTCOMES:
Subjective and objective International Knee Documentation Committee | Two years
  Clinical scores widely used to assess knee function and symptoms Values: 0 (worst score) to 100 (best score) for subjective IKDC; A (best score)-B-C-D (worst score) for objective IKDC (International Knee Documentation Committee)
VAS pain | Two years
  Numerical score to quantitatively assess the intensity of pain (0-10)
Kellgreen-Lawrence | Two years
  Radiographical score that graded knee ostheoarthritis
Knee Laxity | Two years
  Assessment of knee anterior posterior laxity and quantification of Pivot shift using measurement devices (KT-1000; Kira)
Failure and complications | Two years
  Failures and complication rate for each arm of the study

SECONDARY OUTCOMES:
Short Form-36 Health Survey | Two years
  SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting and are now widely utilized by managed care organizations and by Medicare for routine monitoring and assessment of care outcomes in adult patients.
Anterior knee pain | Two years
  The patients will report in dicotomic way (yes/no) the presence/absence of pain referred to patello-femural joint.
Global satisfaction about the surgical procedure | Two years
  The patients will report in dicotomic way (yes/no) if they are satisfied with the surgical procedure results
Tight circumference | Two years
  Tight circumference measured 5 cm and 15 cm above the patella; it is a direct measurement of quadriceps trophism and indirectly explore the muscular status of affected limb.
Lysholm knee scoring scale | Two years
  Clinical score used to assess knee function in context of ligamentary and meniscal lesions Values: 0 (worst score) to 100 (best score)
Tegner activity scale | Two years
  Score that graded activity based on work and sports referred to knee status Values: 0 (worst score) to 10 (best score)

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Zaffagnini, MD Prof, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

REFERENCES:
- [Background] Samuelsen BT, Webster KE, Johnson NR, Hewett TE, Krych AJ. Hamstring Autograft versus Patellar Tendon Autograft for ACL Reconstruction: Is There a Difference in Graft Failure Rate? A Meta-analysis of 47,613 Patients. Clin Orthop Relat Res. 2017 Oct;475(10):2459-2468. doi: 10.1007/s11999-017-5278-9. PMID 28205075
- [Background] Getgood A, Hewison C, Bryant D, Litchfield R, Heard M, Buchko G, Hiemstra LA, Willits KR, Firth A, MacDonald P; Stability Study Group. No Difference in Functional Outcomes When Lateral Extra-Articular Tenodesis Is Added to Anterior Cruciate Ligament Reconstruction in Young Active Patients: The Stability Study. Arthroscopy. 2020 Jun;36(6):1690-1701. doi: 10.1016/j.arthro.2020.02.015. Epub 2020 Mar 6. PMID 32147485
- [Background] Zaffagnini S, Marcheggiani Muccioli GM, Grassi A, Roberti di Sarsina T, Raggi F, Signorelli C, Urrizola F, Spinnato P, Rimondi E, Marcacci M. Over-the-top ACL Reconstruction Plus Extra-articular Lateral Tenodesis With Hamstring Tendon Grafts: Prospective Evaluation With 20-Year Minimum Follow-up. Am J Sports Med. 2017 Dec;45(14):3233-3242. doi: 10.1177/0363546517723013. Epub 2017 Sep 18. PMID 28922015
- [Background] Xie X, Xiao Z, Li Q, Zhu B, Chen J, Chen H, Yang F, Chen Y, Lai Q, Liu X. Increased incidence of osteoarthritis of knee joint after ACL reconstruction with bone-patellar tendon-bone autografts than hamstring autografts: a meta-analysis of 1,443 patients at a minimum of 5 years. Eur J Orthop Surg Traumatol. 2015 Jan;25(1):149-59. doi: 10.1007/s00590-014-1459-3. Epub 2014 Apr 21. PMID 24748500
- [Background] Mouarbes D, Menetrey J, Marot V, Courtot L, Berard E, Cavaignac E. Anterior Cruciate Ligament Reconstruction: A Systematic Review and Meta-analysis of Outcomes for Quadriceps Tendon Autograft Versus Bone-Patellar Tendon-Bone and Hamstring-Tendon Autografts. Am J Sports Med. 2019 Dec;47(14):3531-3540. doi: 10.1177/0363546518825340. Epub 2019 Feb 21. PMID 30790526
- [Background] Chen H, Liu H, Chen L. Patellar Tendon Versus 4-Strand Semitendinosus and Gracilis Autografts for Anterior Cruciate Ligament Reconstruction: A Meta-analysis of Randomized Controlled Trials With Mid- to Long-Term Follow-Up. Arthroscopy. 2020 Aug;36(8):2279-2291.e8. doi: 10.1016/j.arthro.2020.04.024. Epub 2020 May 7. PMID 32387652
- [Background] Curado J, Hulet C, Hardy P, Jenny JY, Rousseau R, Lucet A, Steltzlen C, Morin V, Grimaud O, Bouguennec N, Pujol N, Sonnery-Cottet B, Graveleau N; French Society for Orthopaedic, Trauma Surgery (Societe francaise de chirurgie orthopedique et traumatologique, SoFCOT). Very long-term osteoarthritis rate after anterior cruciate ligament reconstruction: 182 cases with 22-year' follow-up. Orthop Traumatol Surg Res. 2020 May;106(3):459-463. doi: 10.1016/j.otsr.2019.09.034. Epub 2020 Feb 1. PMID 32019734
- [Result] Zaffagnini S, Marcacci M, Lo Presti M, Giordano G, Iacono F, Neri MP. Prospective and randomized evaluation of ACL reconstruction with three techniques: a clinical and radiographic evaluation at 5 years follow-up. Knee Surg Sports Traumatol Arthrosc. 2006 Nov;14(11):1060-9. doi: 10.1007/s00167-006-0130-x. Epub 2006 Aug 15. PMID 16909301